CLINICAL TRIAL: NCT02665546
Title: Evaluation of Exercise Capacity and Mechanisms of Exercise Limitation in Patients With Pulmonary Langerhans Cell Histiocytosis
Brief Title: Evaluation of Exercise Capacity and Exercise Limitation in Patients With Pulmonary Langerhans Cell Histiocytosis
Status: Completed | Type: Observational
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Bruno Guedes Baldi, phD, InCor Heart Institute
Other Study IDs: 4275/15/102
Record Dates: First submitted 2016-01-14; First posted 2016-01-27 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Dyspnea; pulmonary hypertension; Histiocytosis Langerhans cells; exercise test
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Dyspnea; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Patients with diagnosis of LCH based on histopathological or clinical and radiological findings.
- Controls: Current or ex smokers matched with cases for age, gender and smoking history.

SUMMARY:
Pulmonary Langerhans Histiocytosis Cells (PLCH) is characterized by infiltration of Langerhans cells and formation of loose granulomas with lymphocytic infiltrate and formation of nodular and cystic lesions on chest CT, and is often associated with smoking. Functionally, there may be obstructive and / or restrictive defect, with reduced carbon monoxide diffusing capacity. Dyspnea and lower exercise tolerance are common in PLCH, but exercise capacity in this disease is poorly understood and has not been compared to controls. Besides, the mechanisms involved in limiting exercise are poorly understood and cover multiple factors such as change in gas exchange, pulmonary hypertension (PH), dynamic hyperinflation, physical deconditioning and left heart failure. The involvement of pulmonary circulation in PLCH has unknown prevalence, but contributes to the symptoms. In the PH classification, PLCH belongs to the group 5, of multifactorial etiology. The definition of the presence and contribution of dyspnea mechanisms in different severities of PLCH is important to understanding the disease and individualization of treatment. The objective of the study is to evaluate the exercise capacity of patients with HCLP, and determinate mechanisms of dyspnea and lower exercise tolerance beyond its impact on quality of life.

DETAILED DESCRIPTION:
Langerhans cells are antigen-presenting cells of monocyte-macrophage lineage present in various epithelium like airways. Langerhans cell histiocytosis (LCH), also called histiocytosis X or pulmonary eosinophilic granulomatosis, are characterized by proliferation and infiltration of Langerhans cells in the affected organs, including skin, lung, bones, pituitary gland, liver, lymph nodes and thyroid gland.

Several clinical presentations have been described. In the pediatric population, clonal neoplastic processes are responsible for acute disseminated forms (Letterer-Siwe syndrome) or multifocal forms (Syndrome Hand-Schuller-Christian),and both have an unfavorable prognosis.

In adults, LCH may affect one or several organs in a multisystemic disease. The pulmonary form is usually sporadic and occurs almost exclusively in smokers, with smoking history of at least 20 pack-years. It is believed that, unlike systemic forms, exposure to tobacco antigens generates a polyclonal response with recruitment and accumulation of Langerhans cells throughout the interstitium of small airways.

LCH is a rare condition. The prevalence of 3.4% found in a series of 502 surgical lung biopsies may be underestimated, because many patients may improve spontaneously or may be asymptomatic and diagnosis is defined based on radiological findings. The main clinical features are cough, dyspnea and respiratory failure. The mean age of diagnosis is between 20 and 40 years. Men and women are equally affected, which probably reflects the characteristics of smoking habits nowadays.

In the study of Vassallo and colleagues, median survival was 12.5 years between diagnosis and death in patients with LCH, which is lower than that described in general population. Among the predictors of poor prognosis In this study the predictors of worse prognosis include an obstructive pattern, air trapping and reduction in carbon monoxide diffusing capacity (DLCO) in pulmonary function tests.

The diagnosis of pulmonary LCH may be established by the combination of compatible clinical and radiological findings in smoking patients. In high-resolution computed tomography, the typical pattern is the coexistence of cysts and nodules, predominantly in the upper and middle lobes, and tends to spare the basal portions of the lungs. Moreover, interstitial infiltrates, reticular densities and architectural distortion degrees may be found. Computed tomography, such as in others cystic lung diseases, is useful in monitoring the disease progression and to assess treatment response.

In some cases, histopathological examination may be necessary, preferably by surgical biopsy, but transbronchial or transthoracic biopsy may be sufficient in selected patients.

In pathology, LCH presents with focal changes, separated by apparently normal lung parenchyma, and diffuse distribution with bronchiolar predominance and the presence of Langerhans cells organized into loose granulomas and lymphocytic infiltrate.

Lesions of apparently different ages can be found: Initially, eccentric infiltration of the walls of respiratory bronchioles is found, which promotes gradual destruction. Inflammatory cells and Langerhans cells are also present. In advanced disease, lesions are replaced by stellar fibrotic scars bordering cystic spaces of different sizes.

In electron microscopy, Birbeck granules may be identified, which are more numerous in cells associated with the disease than in normal Langerhans cells. The immunohistochemical staining shows membrane antigens on the cell surface of Langerhans cells, such as S100 and CD1a - the latter is more specific - and confirms the diagnosis.

Up to 15% of pulmonary function tests may be normal in patients with LCH. The earliest finding is reduced DLCO. The most frequent changes are airflow obstruction and air trapping. Restriction can be found in more advanced cases. In 102 patients with LCH evaluated by Vassallo and colleagues, mean DLCO was 64% of predicted, and restrictive and obstructive disorders were found in, respectively, 27.2% and 45.7% of all patients.

Smoking cessation is mandatory in the treatment of patients with pulmonary LCH, and this isolated therapy determine partial or complete resolution or stabilization of lesions in the majority of patients. In some patients, corticosteroids and cytotoxic agents, such as cladribine and etoposide, may be necessary. However, there is lack of robust evidence about the benefit of these medications. Lung transplantation should be considered in advanced cases.

Extrapulmonary involvement in LCH occurs in approximately 15% of adults and can affect bones, skin or pituitary, which may cause diabetes insipidus. Pneumothorax is one of the most common complications of pulmonary LCH, which is found in 4-17% of patients. Recurrence of pneumothoraxcan be high, especially if conservative treatment is performed.

Pulmonary vascular involvement associated with LCH has been increasingly discussed and described in the literature. Evidence suggests that its contribution to the pathophysiology is more significant than previously believed. Dauriat and colleagues found the presence of pulmonary hypertension (PH) in 92% of LCH patients evaluated for lung transplantation.

Pulmonary hypertension (PH) consists in the involvement of pulmonary vasculature, in which mean pulmonary artery pressure (Mpap), measured by right heart catheterization at rest, is greater than or equal to 25 mmHg. This criteria may be applied if pulmonary capillary pressure at the end of expiration is less than 15 mmHg. In the second International Symposium on Pulmonary Hypertension, which occurred in Evian (France) in 1998, PH was classified according to pathophysiological basis and divided into five groups: 1 - pulmonary arterial hypertension; 2 - related to left heart disease; 3 - secondary to chronic lung disease or hypoxemia; 4 - chronic pulmonary thromboembolism and 5 - Miscellaneous. This classification had several changes since 1998 until the Fifth Symposium, which occured in 2013 in Nice (France).

LCH is currently included in group 5 of PH, which contain multifactorial etiologies of pulmonary hypertension or those with cause not yet fully elucidated.

However, since LCH presents parenchymal abnormalities, PH in this disease may be secondary to hypoxemia and thus belongs to group 3, in which it is believed that remodeling of the parenchyma and, as a result, hypoxemia determine reduction in the cross-sectional area of the vessels, which promotes increase in pulmonary vascular resistance. This mechanism explains why the vast majority of patients with COPD GOLD IV present with mPAP above 20 mmHg, despite the fact that the progression of PH in these cases is slow, with rates of less than 1 mmHg increase per year. In less than 5% of these patients, mPAP exceeds 40 mmHg, a value from which increases the contribution of the cardiovascular component to exercise limitation. In group 3, the presence of HP is a strong predictor of mortality, which is directly proportional to mPAP. In idiopathic pulmonary fibrosis (IPF), survival is inversely proportional to the values of forced vital capacity.

Vascular changes in distant areas of parenchymal abnormalities typical of LCH suggest that there are other mechanisms involved in the pathophysiology of the disease, which still need to be elucidated. It is believed that the production of inflammatory cytokines and growth factors by activated granulomas cause pulmonary vascular remodeling. Moreover, granulomas can directly infiltrate arteries promoting luminal obstruction, fibrosis and hypertrophy of the intima and media. Fartoukh and colleagues retrospectively evaluated 12 lung biopsies of patients with LCH and found arterial and venular changes, respectively, in 60% and 75%. Veno-occlusive-like disease has been seen in one third of these patients.

In patients with symptoms and limitation to exercise which is not fully explained by parenchymal abnormalities, which means disproportionately low DLCO compared with lung volumes, the predominant component is pulmonary arterial hypertension, group 1, in which benefits of specific therapy are proven. Furthermore, levels of pulmonary artery pressure found in patients with HCL are similar of those found in patients of group 1. mPAP levels are higher in patients with LCH compared with those found in patients with COPD or IPF, who have higher impairment in lung volumes.

Some reports or case series demonstrate symptomatic improvement, and also in survival, in exercise capacity and in parameters of right heart catheterization after using single or combined use of pulmonary vasodilators such as phosphodiesterase inhibitors (tadalafil), endothelin receptor antagonists (bosentan) or analogues of prostacyclin (epoprostenol) in patients with LCH.

Thus, it very important to establish a correct diagnosis and also classification of pulmonary hypertension in order to define appropriate treatment, which may result in an increase in survival and an improvement in quality of life after using specific therapy for patients classified in group 1. On the other hand, side effects and expenses with these medications may be prevented in patients with PH included in group 3, and the main focus should be correction of hypoxemia, and treatment of parenchymal disease. Echocardiography is a safe and cost-effective method of screening for evaluation of PH in these patients.

Data about prevalence of PH in patients with LCH is scarce and previous studies only included patients with advanced disease or who are undergoing evaluation for transplantation. A study that evaluates patients with disease with different severities will certainly contribute to the understanding the influence of vascular and parenchymal components in each patient with LCH.

ELIGIBILITY:
Inclusion Criteria:

* proven diagnosis of pulmonary Langerhans cell histiocytosis based on histopathological or clinical and radiological findings;

Exclusion Criteria:

* lung transplantation
* cognitive or musculoskeletal disorders that preclude exercise test;
* severe or decompensated heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of pulmonary Langerhans cell histiocytosis and current or ex smokers followed at the outpatient clinic of the Pulmonary Division of the Hospital das Clinicas of the University of Sao Paulo
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Maximal O2 uptake capacity (VO2 max) | Baseline
  Maximal O2 uptake capacity (VO2 max) during a cardiopulmonary exercise test (mL/kg/min)

SECONDARY OUTCOMES:
Six-minute walk distance | Baseline
  Distance during a six-minute walk test in meters
Short Form Health Survey (SF-36) | Baseline
  SF-36 questionnaire to evaluate quality of life
Diffusing capacity for carbon monoxide | Baseline
  Diffusing capacity for carbon monoxide (mL/min/mmHg)
Inspiratory capacity | Baseline
  Serial measurement of inspiratory capacity during incremental cardiopulmonary exercise test (L)
Forced expiratory volume in the first 1 second (FEV1) | baseline
  FEV1 (Pulmonary lung function - spirometry) - L
Velocity measurement of tricuspid regurgitant jet | Baseline
  Velocity measurement of tricuspid regurgitant jet evaluated by transthoracic echocardiography (m/s)
Residual volume/total lung capacity ratio | baseline
  Residual volume/total lung capacity ratio evaluated in pulmonary lung function - plethysmography
Residual volume | Baseline
  Residual volume evaluated in pulmonary lung function - plethysmography (L)
Baseline Dyspnea Index | Baseline
  Baseline Dyspnea Index
Six-minute walk test desaturation | Baseline
  Desaturation during a six-minute walk test (%)
Ejection fraction | Baseline
  Ejection fraction evaluated by transthoracic echocardiography (%)
Diameter of the cardiac chambers | Baseline
  Diameter of the cardiac chambers evaluated by transthoracic echocardiography (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno G Baldi, md, PhD, Principal Investigator — InCor Heart Institute
Locations (1):
- InCor Heart Institute, São Paulo, Brazil

REFERENCES:
- [Background] Vassallo R, Ryu JH, Schroeder DR, Decker PA, Limper AH. Clinical outcomes of pulmonary Langerhans'-cell histiocytosis in adults. N Engl J Med. 2002 Feb 14;346(7):484-90. doi: 10.1056/NEJMoa012087. PMID 11844849
- [Background] Torre O, Harari S. The diagnosis of cystic lung diseases: a role for bronchoalveolar lavage and transbronchial biopsy? Respir Med. 2010 Jul;104 Suppl 1:S81-5. doi: 10.1016/j.rmed.2010.03.021. Epub 2010 Apr 28. PMID 20430602
- [Background] Seely JM, Salahudeen S Sr, Cadaval-Goncalves AT, Jamieson DH, Dennie CJ, Matzinger FR, Souza CA. Pulmonary Langerhans cell histiocytosis: a comparative study of computed tomography in children and adults. J Thorac Imaging. 2012 Jan;27(1):65-70. doi: 10.1097/RTI.0b013e3181f49eb6. PMID 21042223
- [Background] Caminati A, Cavazza A, Sverzellati N, Harari S. An integrated approach in the diagnosis of smoking-related interstitial lung diseases. Eur Respir Rev. 2012 Sep 1;21(125):207-17. doi: 10.1183/09059180.00003112. PMID 22941885
- [Background] Attili AK, Kazerooni EA, Gross BH, Flaherty KR, Myers JL, Martinez FJ. Smoking-related interstitial lung disease: radiologic-clinical-pathologic correlation. Radiographics. 2008 Sep-Oct;28(5):1383-96; discussion 1396-8. doi: 10.1148/rg.285075223. PMID 18794314
- [Background] Mason RH, Foley NM, Branley HM, Adamali HI, Hetzel M, Maher TM, Suntharalingam J. Pulmonary Langerhans cell histiocytosis (PLCH): a new UK register. Thorax. 2014 Aug;69(8):766-7. doi: 10.1136/thoraxjnl-2013-204313. Epub 2014 Jan 30. PMID 24482091
- [Background] Tazi A. Adult pulmonary Langerhans' cell histiocytosis. Eur Respir J. 2006 Jun;27(6):1272-85. doi: 10.1183/09031936.06.00024004. PMID 16772390
- [Background] Paciocco G, Uslenghi E, Bianchi A, Mazzarella G, Roviaro GC, Vecchi G, Harari S. Diffuse cystic lung diseases: correlation between radiologic and functional status. Chest. 2004 Jan;125(1):135-42. doi: 10.1378/chest.125.1.135. PMID 14718432
- [Background] Fukuda Y, Miura S, Fujimi K, Yano M, Nishikawa H, Yanagisawa J, Hiratsuka M, Shiraishi T, Iwasaki A, Saku K. Effects of treatment with a combination of cardiac rehabilitation and bosentan in patients with pulmonary Langerhans cell histiocytosis associated with pulmonary hypertension. Eur J Prev Cardiol. 2014 Dec;21(12):1481-3. doi: 10.1177/2047487313497603. Epub 2013 Jul 29. PMID 23897898
- [Background] Soler P, Bergeron A, Kambouchner M, Groussard O, Brauner M, Grenier P, Crestani B, Mal H, Tazi A, Battesti JP, Loiseau P, Valeyre D. Is high-resolution computed tomography a reliable tool to predict the histopathological activity of pulmonary Langerhans cell histiocytosis? Am J Respir Crit Care Med. 2000 Jul;162(1):264-70. doi: 10.1164/ajrccm.162.1.9906010. PMID 10903252
- [Background] Ryu JH, Tian X, Baqir M, Xu K. Diffuse cystic lung diseases. Front Med. 2013 Sep;7(3):316-27. doi: 10.1007/s11684-013-0269-z. Epub 2013 May 11. PMID 23666611
- [Background] Fartoukh M, Humbert M, Capron F, Maitre S, Parent F, Le Gall C, Sitbon O, Herve P, Duroux P, Simonneau G. Severe pulmonary hypertension in histiocytosis X. Am J Respir Crit Care Med. 2000 Jan;161(1):216-23. doi: 10.1164/ajrccm.161.1.9807024. PMID 10619823
- [Background] Lorillon G, Bergeron A, Detourmignies L, Jouneau S, Wallaert B, Frija J, Tazi A. Cladribine is effective against cystic pulmonary Langerhans cell histiocytosis. Am J Respir Crit Care Med. 2012 Nov 1;186(9):930-2. doi: 10.1164/ajrccm.186.9.930. No abstract available. PMID 23118088
- [Background] Aerni MR, Aubry MC, Myers JL, Vassallo R. Complete remission of nodular pulmonary Langerhans cell histiocytosis lesions induced by 2-chlorodeoxyadenosine in a non-smoker. Respir Med. 2008 Feb;102(2):316-9. doi: 10.1016/j.rmed.2007.09.002. Epub 2007 Nov 1. PMID 17935961
- [Background] Benyounes B, Crestani B, Couvelard A, Vissuzaine C, Aubier M. Steroid-responsive pulmonary hypertension in a patient with Langerhans' cell granulomatosis (histiocytosis X). Chest. 1996 Jul;110(1):284-6. doi: 10.1378/chest.110.1.284. PMID 8681645
- [Background] Abbritti M, Mazzei MA, Bargagli E, Refini RM, Penza F, Perari MG, Volterrani L, Rottoli P. Utility of spiral CAT scan in the follow-up of patients with pulmonary Langerhans cell histiocytosis. Eur J Radiol. 2012 Aug;81(8):1907-12. doi: 10.1016/j.ejrad.2011.04.018. Epub 2011 May 6. PMID 21549535
- [Background] Mendez JL, Nadrous HF, Vassallo R, Decker PA, Ryu JH. Pneumothorax in pulmonary Langerhans cell histiocytosis. Chest. 2004 Mar;125(3):1028-32. doi: 10.1378/chest.125.3.1028. PMID 15006964
- [Background] Dauriat G, Mal H, Thabut G, Mornex JF, Bertocchi M, Tronc F, Leroy-Ladurie F, Dartevelle P, Reynaud-Gaubert M, Thomas P, Pison C, Blin D, Stern M, Bonnette P, Dromer C, Velly JF, Brugiere O, Leseche G, Fournier M. Lung transplantation for pulmonary langerhans' cell histiocytosis: a multicenter analysis. Transplantation. 2006 Mar 15;81(5):746-50. doi: 10.1097/01.tp.0000200304.64613.af. PMID 16534477
- [Background] Hoeper MM, Bogaard HJ, Condliffe R, Frantz R, Khanna D, Kurzyna M, Langleben D, Manes A, Satoh T, Torres F, Wilkins MR, Badesch DB. Definitions and diagnosis of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D42-50. doi: 10.1016/j.jacc.2013.10.032. PMID 24355641
- [Background] Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT); Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G. Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2009 Dec;34(6):1219-63. doi: 10.1183/09031936.00139009. Epub 2009 Sep 12. No abstract available. PMID 19749199
- [Background] Seeger W, Adir Y, Barbera JA, Champion H, Coghlan JG, Cottin V, De Marco T, Galie N, Ghio S, Gibbs S, Martinez FJ, Semigran MJ, Simonneau G, Wells AU, Vachiery JL. Pulmonary hypertension in chronic lung diseases. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D109-16. doi: 10.1016/j.jacc.2013.10.036. PMID 24355635
- [Background] Le Pavec J, Lorillon G, Jais X, Tcherakian C, Feuillet S, Dorfmuller P, Simonneau G, Humbert M, Tazi A. Pulmonary Langerhans cell histiocytosis-associated pulmonary hypertension: clinical characteristics and impact of pulmonary arterial hypertension therapies. Chest. 2012 Nov;142(5):1150-1157. doi: 10.1378/chest.11-2490. PMID 22459770
- [Background] Kiakouama L, Cottin V, Etienne-Mastroianni B, Khouatra C, Humbert M, Cordier JF. Severe pulmonary hypertension in histiocytosis X: long-term improvement with bosentan. Eur Respir J. 2010 Jul;36(1):202-4. doi: 10.1183/09031936.00004810. No abstract available. PMID 20595165
- [Background] Bendayan D, Shitrit D, Kramer MR. Combination therapy with prostacyclin and tadalafil for severe pulmonary arterial hypertension: a pilot study. Respirology. 2008 Nov;13(6):916-8. doi: 10.1111/j.1440-1843.2007.01176.x. PMID 18811891
- [Derived] Heiden GI, Sobral JB, Freitas CSG, Pereira de Albuquerque AL, Salge JM, Kairalla RA, Fernandes CJCDS, Carvalho CRR, Souza R, Baldi BG. Mechanisms of Exercise Limitation and Prevalence of Pulmonary Hypertension in Pulmonary Langerhans Cell Histiocytosis. Chest. 2020 Dec;158(6):2440-2448. doi: 10.1016/j.chest.2020.05.609. Epub 2020 Jun 29. PMID 32615192